CLINICAL TRIAL: NCT02269969
Title: Once Daily Aminoglycoside Pharmacokinetics and Optimal Dosing in the Burn Population: A Prospective Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sandra Walker (Other)
Responsible Party: Sponsor-Investigator, Sandra Walker, Clinician Scientist, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 183-2014
Record Dates: First submitted 2014-10-08; First posted 2014-10-21 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Burns; Infection
Keywords: Aminoglycoside; Pharmacokinetics; Once daily dosing
MeSH Terms: conditions — Burns; Infections | interventions — Tobramycin

ARMS (1):
- Once daily aminoglycoside (Experimental): Once daily dosing of Tobramycin
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Tobramycin

SUMMARY:
Effective antimicrobial use in the burn population is important since this population is at an increased risk for infections during their stay in hospital as a result of their burn injury. Tobramycin is an antibiotic that has activity against common burn wound associated pathogens, such as Pseudomonas Aeruginosa, and its use is becoming increasingly relevant due to the increased incidence of bacterial resistance to currently utilized antibiotics. Once daily dosing of tobramycin has been safely and effectively used in the majority of infected patients for many years with the proposed benefits of optimized antibacterial activity and reduced nephrotoxicity compared to traditional dosing. But, the once daily dosing regimen has yet to be validated in the burn population. The purpose of this study is to validate the plausibility of once daily tobramycin dosing in the burn population with intent to determine a safe, effective, and efficient dosing regimen for this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult burn patient (≥ 18 years old)
* Total burn surface area less than 20%
* At least 48 hours after the time of the initial burn injury event
* Has a suspected or confirmed infection
* Has been receiving antibiotic therapy for at least 24 hours

Exclusion Criteria:

* Pediatric patients (< 18 years old);
* Pregnant
* Documented history of cochlear or vestibular injury
* Creatinine clearance < 50 ml/min
* Requiring any modality of dialysis
* Has been receiving antibiotic therapy for longer than 72 hours
* Known allergy or adverse reaction to aminoglycoside antibiotics
* Known allergy or adverse reaction to sulfites
* Diagnosis of Parkinson's disease or myasthenia gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients able to achieve therapeutic target | 24 hours
Clearance of tobramycin in the burn population | 24 hours
Volume of distribution of tobramycin in the burn population | 24 hours
Breakpoint in tobramycin clearance based on time post-burn, body burn surface area, inhalation injury score, or percentage of open wounds | 24 hours
Breakpoint in tobramycin volume of distribution based on time post-burn, body burn surface area, inhalation injury score, or percentage of open wounds | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada